CLINICAL TRIAL: NCT06591247
Title: Evaluation of Stripping for Cervical Ripening - A Randomized Controlled Study
Brief Title: Membrane Stripping for Cervical Ripening
Acronym: Stripping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Gal Cohen, Gal Cohen MD, Principal Investigator, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0067-23-MMC
Record Dates: First submitted 2024-08-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Labor, Induced; Cervical Ripening; Balloon Induction; Membrane Stripping; Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Balloon Catheter induction (Active Comparator): A Double balloon catheter will be inserted for 12 hours in this group of women
  Interventions: Device: Double Baloon Catheter
- Membrane stripping (Active Comparator): This group of women will undergo membrane stripping twice (every 4-6 hours) over a period of 12 hours
  Interventions: Procedure: Membrane Stripping

INTERVENTIONS:
Device: Double Baloon Catheter — A double Baloon Catheter will be inserted for 12 hours to one of the arms of the study
  Arms: Double Balloon Catheter induction
Procedure: Membrane Stripping — Stripping will be considered as 3-5 rotations of separating the amniotic sac from the cervix and will be perfomed twice (every 4-6 hours)
  Arms: Membrane stripping

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of membrane stripping in cervical ripening compared to double balloon catheter induction.

The study population consists of women undergoing labor induction.

The main questions it aims to answer are:

1. Is membrane stripping as effective as double balloon catheter induction in cervical ripening?
2. What is the influence of membrane stripping on the time required for cervical ripening, delivery duration, and maternal and fetal outcomes compared to balloon induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above
* Patients with a cervical dilation of at least 1 cm
* Full-term pregnancy
* Cephalic presentation
* No contraindication to vaginal delivery

Exclusion Criteria:

* Patients with rupture of membranes
* Patients who do not require cervical ripening and proceed directly to the delivery room for induction with oxytocin
* Patients for whom the use of a double-balloon catheter is contraindicated
* Twin pregnancies
* Pregnancies with macrosomic fetuses where vaginal delivery is contraindicated
* Vaginal deliveries after a cesarean section
* Patients with maternal or fetal pathologies that do not allow for vaginal delivery due to concerns about fetal or maternal distress

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of successful cervical ripening at the end of 12 hours, duration of cervical ripening | from 12 hours after intervention until patient&s discharge or 150 hours, whichever came first, assessed up to 100 months
  What percentage of the women in this arm had a successful cervical ripening after 12 hours

SECONDARY OUTCOMES:
Rates of vaginal delivery within 24 hours | from 12 hours after intervention until patients discharge or 150 hours, whichever came first, assessed up to 100 months
  What percentage of the women in this arm delivered within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Central District, Israel